CLINICAL TRIAL: NCT02279043
Title: Peer Influence on Intrauterine Contraceptive Behavior and Attitudes in an Online Social Community
Brief Title: Online Peer Influence on IUD Behaviors and Attitudes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: William and Flora Hewlett Foundation (Other); University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Christine Dehlendorf, Associate Professor, School of Medicine, Department of Family and Community Medicine, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2014-9716; 820383 (Other: University of Pennsylvania Institutional Review Board); 14-14827 (Other: UCSF Committee on Human Research)
Record Dates: First submitted 2014-10-27; First posted 2014-10-30 (Estimated); Results first posted 2019-03-11 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Contraception
Keywords: IUD; IUC; birth control; contraception; online
MeSH Terms: interventions — Drug Interactions

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Intervention (Experimental): IUC users and non-IUC user participants randomized to the intervention arm will take part in small intervention groups in an online community called Birth Control Connect for twelve days. There will be up to 35 intervention groups with 9 members each. Non-IUC users in these groups will receive the intervention of Interaction with users of IUC and non-IUC users in the context of the online community. About 50% of participants in intervention groups will be current IUC users, and 50% will not be current IUC users. We will measure the attitudes and behaviors of those who do not have IUC before and after the intervention, considering social exposure to IUC users as a possible predictor of changes in knowledge, attitude and behavior.
  Interventions: Behavioral: Interaction with users of IUC and non-IUC users
- Control (Placebo Comparator): Participants randomized to the control arm will take part in Birth Control Connect control groups identical to those in the intervention arm, except no participants in the control arm will be current IUC users. Therefore, participants in the control arm will have interaction with non-IUC users only. We will measure these participants' attitudes and behavior related to IUC use before and after the twelve-day study period, and compare results to those of participants in the intervention arm. There will be up to 35 control groups of 9 members each.
  Interventions: Behavioral: Interaction with non-IUC users only
- IUC users (No Intervention): IUC users will be recruited to populate intervention groups. Interaction with IUC users will be the intervention for non-IUC users randomized to the intervention arm. IUC users will receive no intervention.

INTERVENTIONS:
Behavioral: Interaction with users of IUC and non-IUC users — Birth Control Connect is an online community where women will be invited to share their personal experiences with birth control. Birth Control Connect group sessions will last for twelve days. Each day, participants will be prompted to respond to questions in the group (e.g. "If you're using a birth control method right now, how did you choose it?"). Participants will also be able to pose questions to other members of the group and respond to other members' questions. Half of participants in Birth Control Connect intervention groups will be current IUC users.
  Arms: Intervention
Behavioral: Interaction with non-IUC users only — Birth Control Connect is an online community where women will be invited to share their personal experiences with birth control. Birth Control Connect group sessions will last for twelve days. Each day, participants will be prompted to respond to questions in the group (e.g. "If you're using a birth control method right now, how did you choose it?"). Participants will also be able to pose questions to other members of the group and respond to other members' questions.
  Arms: Control

SUMMARY:
This study will look at women's social communication about IUDs (intrauterine devices) and their attitudes and behavior related to IUD use. The researchers will design an online community where women can talk to each other about their experiences with birth control. We will examine whether social exposure to IUD users in this setting is associated with change in attitudes and behavior among women who have never had an IUD.

DETAILED DESCRIPTION:
Study Design:

University of Pennsylvania researchers will conduct a randomized controlled trial to examine whether there is an association between social exposure to women who use intrauterine contraception (IUC) as their method of birth control and change in IUC attitudes and behavior among women who have never used IUC. The intervention used to test this association will be an online social community, designed by the researchers, in which women will be invited to share their personal experiences with birth control methods they have used. Non-IUC user participants will be randomized to either the intervention or control conditions. The intervention condition will consist of small online social groups in which non-IUC user participants will interact with IUC user participants. The control condition will consist of online groups identical to intervention groups, except that no IUC user participants will be in these groups. Participants will interact within small groups for twelve days each. Non-IUC user participants will complete surveys before and after the twelve-day intervention that measure IUC attitudes and behavior. UCSF researchers will conduct analysis on deidentified data obtained from this study.

Hypothesis:

It is hypothesized that among women who have never used IUC, there is an association between social exposure to IUC users and change in attitudes and behavior related to IUC use. It is also hypothesized that exposure to IUC users is associated with positive change in knowledge of IUC use and efficacy and positive change in IUC-related information-seeking.

Aims:

The study has three aims:

Aim 1: To determine whether exposure to IUC users in an online community is associated with change in women's attitudes and behavior related to IUC use.

Aim 2: To determine whether an association between exposure to IUC users and change in women's IUC attitudes and behavior varies by women's race/ethnicity.

Aim 3: To observe the content of women's interactions about IUC and other birth control methods in an online social community.

Data analysis:

In order to address Aim 1, we will first conduct univariate analysis and obtain descriptive statistics (including mean, median, mode, variance, and range) on demographic characteristics and IUC attitudes and behaviors among participants in the intervention and control groups. In bivariate analysis, we will use chi-square tests to examine the relationship between study condition and IUC-related behaviors, as measured on the post-survey. We will use t-tests to examine relationships between condition and post-survey IUC attitudes, and matched t-tests to examine the relationships between conditions and changes in IUC attitudes. If data on attitudes is not normally distributed, we will use the appropriate non-parametric tests instead of t-tests.

We will conduct multivariate analyses for those outcomes associated with intervention condition in bivariate tests. Multivariate analysis for Aim 1 will include mixed-effects regression to examine associations at both the individual and cluster levels. We will use multiple linear regression for continuous outcomes and multiple logistic regression for binary outcomes. Regression models will test associations between intervention and control conditions and outcome IUC attitude and behavior variables. We will obtain regression coefficients from linear regression models and odds ratios from logistic regression models in order to describe the associations between study arms and outcomes.

In order to address Aim 2, we will examine bivariate relationships between the racial/ethnic categories of participants and outcome attitude and behavior variables, using chi-square tests for binary outcomes and t-tests or appropriate non-parametric tests for continuous outcomes. We will use multiple linear and/or logistic regression to test possible associations between race/ethnicity and outcome variables, controlling for other background variables. Resulting regression coefficients and odds ratios will describe whether the effect of the intervention was greater for women in some racial/ethnic groups as compared to others.

In order to address Aim 3, we will perform qualitative analysis of conversations that take place among group members in the online social groups, using grounded theory methodology. We will examine qualitative data from both the intervention and control groups.

Privacy:

Recruitment and participation in the study will occur online. Participants will only interact with the study from remote locations, so they will not be seen entering or leaving any location affiliated with the study, or interacting with any study personnel. Once registered in the study, participants will only be contacted via secure email that does not indicate the nature of the study in the subject line. The study website will be password-protected to prohibit access to Internet users not participating in the study. Participants' screen names on the site will not contain their real names, and they will not be identifiable to other study participants.

There is minimal risk of privacy loss. Study participants may not want others to know about their interest in or use of birth control, and may have feelings of embarrassment or shame in the event of a loss of study privacy. Additionally, birth control use may be a sensitive topic in the personal relationships of some study participants, and a loss of privacy could lead to strain or conflict in these personal relationships.

Confidentiality:

Data collected by researchers at the University of Pennsylvania will be stored on a secure network at their site. Only University of Pennsylvania study staff will have access to data on this network. University of PEnnsylvania staff will remove all identifiers from the data and export the data to researchers at UCSF via secure email. Deidentified data will be stored at on a secure UCSF server. Only the study staff will have access to the data, and we will not have access to the key.

ELIGIBILITY:
Inclusion Criteria:

Non-IUC users:

* Women
* Age 18 - 45
* Sexually active with men
* Do not want to get pregnant in the next year
* Want to learn more about different birth control methods

IUC users

* Women
* Age 18-45
* Currently uses IUC (Paragard, Mirena, or Skyla)

Exclusion Criteria:

Non-IUC users

* Previous IUC use
* Not able to become pregnant

IUC users

-Using IUC for other reason, and not pregnancy prevention

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 630 (Actual)
Dates: Start 2015-10; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Damon Centola, PhD, Principal Investigator — University of Pennsylvania, Annenberg School of Communication; Christine Dehlendorf, MD, MAS, Principal Investigator — University of California, San Francisco
Locations (1):
- University of Pennsylvania, Annenberg School of Communication, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Deidentified data will be shared with UCSF researchers through secure email.

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: IUC users and non-IUC user participants randomized to the intervention arm will take part in small intervention groups in an online community called Birth Control Connect for twelve days. There will be up to 35 intervention groups with 9 members each. Non-IUC users in these groups will receive the intervention of Interaction with users of IUC and non-IUC users in the context of the online community. About 50% of participants in intervention groups will be current IUC users, and 50% will not be current IUC users.
  Interaction with users of IUC and non-IUC users: Birth Control Connect group sessions will last for twelve days. Each day, participants will be prompted to respond to questions in the group. Participants will also be able to pose questions to other members of the group and respond to other members' questions. Half of participants in Birth Control Connect intervention groups will be current IUC users.
- Control: Participants randomized to the control arm will take part in Birth Control Connect control groups identical to those in the intervention arm, except no participants in the control arm will be current IUC users. Therefore, participants in the control arm will have interaction with non-IUC users only. There will be up to 35 control groups of 9 members each.
  Interaction with non-IUC users only: Birth Control Connect group sessions will last for twelve days. Each day, participants will be prompted to respond to questions in the group (e.g. "If you're using a birth control method right now, how did you choose it?"). Participants will also be able to pose questions to other members of the group and respond to other members' questions.
Period: Overall Study
Arm/Group | Intervention | Control | IUC Users
Started | 175 | 315 | 140
Completed | 128 | 226 | 140
Not Completed | 47 | 89 | 0
Not completed — Post-rand. exclusion - not eligible | 1 | 1 | 0
Not completed — Lost to Follow-up | 46 | 88 | 0

BASELINE CHARACTERISTICS:
Population: Data analyzed for non-IUC user participants only, not IUC users. Post-randomization excluded participants (n=2) not included in baseline analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | IUC Users | Total
Number analyzed (Participants) | 174 | 314 | 0 | 488
Age, Customized [Count of Participants; unit: Participants]
  18-24 | 90 | 159 |  | 249
  25-34 | 79 | 137 |  | 216
  35-45 | 5 | 17 |  | 22
  Missing | 0 | 1 |  | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 174 | 314 |  | 488
  Male | 0 | 0 |  | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 12 | 24 |  | 36
  Black/African American | 22 | 38 |  | 60
  Hispanic/Latina | 11 | 36 |  | 47
  White | 116 | 185 |  | 301
  Other | 9 | 18 |  | 27
  Missing | 4 | 13 |  | 17
Number of pregnancies [Count of Participants; unit: Participants]
  0 pregnancies | 82 | 159 |  | 241
  1 or more pregnancies | 21 | 29 |  | 50
  Missing | 71 | 126 |  | 197
Number of children [Count of Participants; unit: Participants]
  0 children | 154 | 282 |  | 436
  1 or more children | 20 | 31 |  | 51
  Missing | 0 | 1 |  | 1
Birth control method used at baseline [Count of Participants; unit: Participants]
  Pill | 95 | 171 |  | 266
  Patch | 2 | 11 |  | 13
  Ring | 10 | 13 |  | 23
  Shot | 12 | 12 |  | 24
  Arm implant | 17 | 29 |  | 46
  Condoms | 64 | 110 |  | 174
  Withdrawal | 37 | 70 |  | 107
  Female sterilization | 4 | 4 |  | 8
  Male sterilization | 2 | 7 |  | 9
  Other | 2 | 6 |  | 8
  None | 7 | 16 |  | 23
Parental education [Count of Participants; unit: Participants]
  High school graduate or less | 31 | 51 |  | 82
  Some college or 4-year college graduate | 56 | 122 |  | 178
  More than 4-year college graduate | 41 | 53 |  | 94
  Missing | 46 | 88 |  | 134

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting IUC Use
Description: Self-reported use of IUC in post-survey
Time Frame: 12 days post-baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 128 | 226
Participants | 2 | 4
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.89, Regression, Logistic; Odds Ratio (OR) = 0.88, 95% CI 2-sided [0.16 to 4.88]

2. Secondary Outcome: Mean Change in Attitude About Hormonal IUC as Method for Self Between Pre-survey and Post-survey
Description: Mean difference of responses to scale in pre- and post-surveys asking participants to rate hormonal IUC as a contraceptive method for themselves, with 0=terrible method and 10=great method
Time Frame: 12 days post-baseline
Population: Number analyzed is less than what is pictured in participant flow diagram because analysis for this outcome only includes those participants who have complete pre-survey and post-survey data pertaining to this outcome.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 119 | 211
units on a scale | 0.50 [0.01 to 0.98] | 0.16 [-0.22 to 0.53]
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.28, t-test, 2 sided

3. Secondary Outcome: Mean Change in Attitude About Hormonal IUC as Method for Women in General Between Pre-survey and Post-survey
Description: Responses to scale in pre- and post-surveys asking participants to rate hormonal IUC as a contraceptive method for women in general, with 0=terrible method and 10=great method
Time Frame: 12 days post-baseline
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 119 | 211
units on a scale | 0.65 [0.25 to 1.04] | 0.05 [-0.27 to 0.38]
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.03, t-test, 2 sided
Statistical Analysis 2: Comparison: Intervention vs Control; Multivariate analysis adjusting for cluster, as association was significant in bivariate test; Test type: Superiority; p = 0.02, Regression, Linear; Slope = 0.59, 95% CI 2-sided [0.08 to 1.11]

4. Secondary Outcome: Mean Change in Attitude About Non-hormonal IUC as Method for Self Between Pre-survey and Post-survey
Description: Responses to scale in pre- and post-surveys asking participants to rate non-hormonal IUC as a contraceptive method for themselves, with 0=terrible method and 10=great method
Time Frame: 12 days post-baseline
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 114 | 207
units on a scale | 0.22 [-0.33 to 0.41] | 0.04 [-0.34 to 0.40]
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.59, t-test, 2 sided

5. Secondary Outcome: Mean Change in Attitude About Non-hormonal IUC as Method for Women in General Between Pre-survey and Post-survey
Description: Responses to scale in pre- and post-surveys asking participants to rate non-hormonal IUC as a contraceptive method for women in general, with 0=terrible method and 10=great method
Time Frame: 12 days post-baseline
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 114 | 211
units on a scale | 0.50 [0.08 to 0.92] | 0 [-0.34 to 0.34]
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.08, t-test, 2 sided

6. Secondary Outcome: Number of Participants With Responses Indicating Knowledge of IUC Safety
Description: Response on 5-point Likert scale of agreement in post-survey on IUC safety. Dichotomized as 4 or 5 (Agree or strongly agree) vs. 1, 2, or 3 (Strongly disagree, disagree, or neither agree nor disagree). Outcome is count of participants responding 4 or 5.
Time Frame: 12 days post-baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 128 | 226
Participants | 103 | 172
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.34, Regression, Logistic; Odds Ratio (OR) = 1.29, 95% CI 2-sided [0.75 to 2.20]

7. Secondary Outcome: Number of Participants With Responses Indicating Knowledge of IUC Effectiveness
Description: Response on 5-point Likert scale of agreement in post-survey on IUC effectiveness. Dichotomized as 4 or 5 (Agree or strongly agree) vs. 1, 2, or 3 (Strongly disagree, disagree, or neither agree nor disagree). Outcome is count of participants responding 4 or 5.
Time Frame: 12 days post-baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 128 | 226
Participants | 115 | 203
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.99, Regression, Logistic; Odds Ratio (OR) = 1.00, 95% CI 2-sided [0.49 to 2.05]

8. Secondary Outcome: Number of Participants With Responses Indicating Knowledge of IUC Being More Effective Than Birth Control Pill
Description: Correct response to post-survey item asking whether IUC is more, less, or as effective as the birth control pill (correct response: more effective).
Time Frame: 12 days post-baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 128 | 226
Participants | 72 | 105
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.08, Regression, Logistic; Odds Ratio (OR) = 1.48, 95% CI 2-sided [0.95 to 2.29]

9. Secondary Outcome: Number of Participants Reporting Informational Support (Receiving New Information From Birth Control Connect)
Description: Response on 5-point Likert scale of agreement in post-survey on whether Birth Control Connect group gave participants information on IUC they didn't have before. Dichotomized as 4 or 5 (Agree or strongly agree) vs. 1, 2, or 3 (Strongly disagree, disagree, or neither agree nor disagree). Outcome is count of participants responding 4 or 5.
Time Frame: 12 days post-baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 128 | 226
Participants | 81 | 116
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.03, Regression, Logistic; Odds Ratio (OR) = 1.63, 95% CI 2-sided [1.05 to 2.58]
Statistical Analysis 2: Comparison: Intervention vs Control; Multivariate analysis adjusting for cluster, as association was significant in bivariate test; Test type: Superiority; p = 0.03, Mixed Models Analysis; Mixed effects logistic regression; Slope = 0.50, 95% CI 2-sided [0.04 to 0.97]

10. Secondary Outcome: Number of Participants Reporting Informational Support (Better Idea of What IUC Would be Like)
Description: Response on 5-point Likert scale of agreement in post-survey on whether Birth Control Connect gave them a better idea of what using IUC would be like. Dichotomized as 4 or 5 (Agree or strongly agree) vs. 1, 2, or 3 (Strongly disagree, disagree, or neither agree nor disagree). Outcome is count of participants responding 4 or 5.
Time Frame: 12 days post-baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 128 | 226
Participants | 90 | 116
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p < 0.01, Regression, Logistic; Odds Ratio (OR) = 2.25, 95% CI 2-sided [1.42 to 3.56]
Statistical Analysis 2: Comparison: Intervention vs Control; Multivariate analysis adjusting for cluster, as association was significant in bivariate test; Test type: Superiority; p < 0.01, Mixed Models Analysis; Mixed effects logistic regression; Slope = 0.84, 95% CI 2-sided [0.33 to 1.35]

11. Secondary Outcome: Number of Participants Reporting Information-seeking on Internet
Description: Report (Yes/No) in post-survey of whether participant had looked on the Internet (outside of Birth Control Connect) for information on IUC since study start. Outcome is count of participants reporting yes.
Time Frame: 12 days post-baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 128 | 226
Participants | 59 | 103
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.93, Regression, Logistic; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.52 to 2.74]

12. Secondary Outcome: Number of Participants Reporting Information-seeking From a Health Care Provider
Description: Report (Yes/No) in post-survey of whether participant had consulted a health care provider about IUC since study start. Outcome is count of participants reporting yes.
Time Frame: 12 days post-baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 128 | 226
Participants | 10 | 15
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.68, Regression, Logistic; Odds Ratio (OR) = 1.19, 95% CI 2-sided [0.52 to 2.74]

13. Secondary Outcome: Number of Participants Reporting Information-seeking From Peers
Description: Report (Yes/No) in post-survey of whether participant had talked to women they know about IUC since study start. Outcome is count of participants reporting yes.
Time Frame: 12 days post-baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 128 | 226
Participants | 56 | 87
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.33, Regression, Logistic; Odds Ratio (OR) = 1.24, 95% CI 2-sided [0.08 to 1.93]

ADVERSE EVENTS:
Time Frame: 12 days post-baseline
Groups:
- Intervention: IUC users and non-IUC user participants randomized to the intervention arm will take part in small intervention groups in an online community called Birth Control Connect for twelve days. There will be up to 35 intervention groups with 9 members each. Non-IUC users in these groups will receive the intervention of interaction with IUC users in the context of the online community.
- Control: Participants randomized to the control arm will take part in Birth Control Connect control groups identical to those in the intervention arm, except no participants in the control arm will be current IUC users. Therefore, participants in the control arm will not have social exposure to IUC users. We will measure these participants' attitudes and behavior related to IUC use before and after the twelve-day study period, and compare results to those of participants in the intervention arm. There will be up to 35 control groups of 9 members each.
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/175 | 0/315
Serious Adverse Events (participants affected / at risk) | 0/175 | 0/315
Other Adverse Events (participants affected / at risk) | 0/175 | 0/315

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No